CLINICAL TRIAL: NCT04028830
Title: Impact on Antibiotic Prescriptions of a Bundle Intervention Conducted by Medical Representatives in General Practitioner Facilities, Based on Operational Demonstration of an Internet Decision Support Tool: Antibioclic
Acronym: ACTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC19_0459
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Antibiotic Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Medical representative presentation with the help internet tool for decision ANTIBIOCLIC
  Interventions: Other: Visit to GPs to promote good antibiotic prescription with the help internet tool for decision: ANTIBIOCLIC
- Arm 2 (Experimental): Medical representative presentation without presentation of the internet tool for decision support
  Interventions: Other: Visit to GPs to promote good antibiotic prescription without presentation of the internet tool for decision support
- Arm 3 (No Intervention): Usual practice without intervention regarding the prescription of antibiotics

INTERVENTIONS:
Other: Visit to GPs to promote good antibiotic prescription with the help internet tool for decision: ANTIBIOCLIC — Visit to GPs to promote good antibiotic prescription with the help internet tool for decision: ANTIBIOCLIC
  Arms: Arm 1
Other: Visit to GPs to promote good antibiotic prescription without presentation of the internet tool for decision support — Visit to GPs to promote good antibiotic prescription without presentation of the internet tool for decision support
  Arms: Arm 2

SUMMARY:
At the international level, several experiments have been conducted to modify antibiotic prescribing practices in GPs. The mere development of training or the mere provision of information on the internet do not seem to change the practices when these interventions are conducted in isolation. On the other hand, various approaches involving communication training, specific educational interventions working on ideas received from examples, interventions at the point of care, and the use of electronic decision support systems have demonstrated beneficial effects on prescription. The fact of sending feedback on their prescribing practices back to GPs also showed an impact

The Antibioclic website was created in 2011. It is an internet tool for prescribing help developed for general practitioners. Every day, it is consulted on average by 9000 health professionals. One question is how far the use of the site makes it possible to modify prescribing practices, which would justify, if need be, to actively promote it to general practitioners who do not use it. (The council of the order of doctors counted a little more than 88000 general practitioners in 2018.)

One challenge would be to implement a strategy:

* combining different actions that have shown their impact: visit to the place of care, awareness of antibiotic resistance, work on preconceived ideas, feedback on practices, use of decision support tools,
* and generalizable nationally.

The proposed study will thus experiment with an intervention modality based on the visit of a medical representative in general practitioner facilities, with:

* antibiotic resistance sensitization,
* work on preconceived ideas,
* feedback on prescriptions,
* use of an Internet tool to assist in the prescription of antibiotics: Antibioclic.

The generalizability of the intervention will be based on the collaboration with the medical representatives , which already intervene in an operational and regular way on this topic on the whole France. The medical representatives, distributed throughout the country, provide regular visits to the GPs and promote good practices. This type of visit to GPs is original internationally, demonstrating its impact on practices is decisive.

The purpose of the research is to compare the effect on antibiotic prescriptions made by general practitioners after 12 months of follow-up, i) an intervention led by the medical representatives in general practitioner facilities, the intervention involving usual visit (antibiotic resistance sensitization, work on preconceived ideas, feedback on practices) and demonstration of the use of Antibioclic, ii) an intervention conducted on the same terms by the the medical representatives but without Antibioclic demonstration, iii) compared to usual practice.

ELIGIBILITY:
Inclusion Criteria:

* GPs practicing on one of the 5 departments of the study having seen at least 100 different patients (whatever the age) during the year preceding the evaluation.

Exclusion Criteria:

* Will not be included attending GPs

  1. who will be identified as having a particular exercise. And / or
  2. that will already be integrated into an antibiotic prevention program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2501 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the overall volume of antibiotics delivered in Defined Daily Dose (DDD) per participating GP, after 12 months of follow-up. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeanmougin P, Larramendy S, Fournier JP, Gaultier A, Rat C. Effect of a Feedback Visit and a Clinical Decision Support System Based on Antibiotic Prescription Audit in Primary Care: Multiarm Cluster-Randomized Controlled Trial. J Med Internet Res. 2024 Dec 18;26:e60535. doi: 10.2196/60535. PMID 39693139